CLINICAL TRIAL: NCT04471675
Title: Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of Albumin-bound Formulation of Docetaxel for Intravenous Infusion in Patients With Advanced Solid Tumors: A Phase 1, Single-center, Open-label, Dose-escalation Study
Brief Title: Evaluation of the Safety and Efficacy of Albumin-bound Docetaxel
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-CSP-001
Record Dates: First submitted 2020-07-07; First posted 2020-07-15 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: solid tumors (Experimental): Albumin-bound docetaxel by intravenous infusion.Patients receive albumin-bound docetaxel once every three weeks (a Cycle), starting at a dose of 50mg/m2.
  Interventions: Drug: Albumin-bound docetaxel

INTERVENTIONS:
Drug: Albumin-bound docetaxel — Albumin-bound docetaxel by intravenous infusion.

SUMMARY:
This trial is an open-label, single-center, dose-escalation and cohort-expansion Phase I clinical study in patients with advanced solid tumors. The aim of this study is designed to evaluate the safety, tolerability, pharmacokinetics and preliminary antitumor activity of albumin-bound formulation of docetaxel for intravenous infusion in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study was conducted in two stages. The first stage (Stage I) is a dose-escalation study. A classic 3+3 design will be used to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D). Patients with advanced solid tumors will be assigned to receive sequentially higher doses of albumin-bound formulation of docetaxel once every three weeks (a Cycle) by intravenous infusion, starting at a dose of 50mg/m2. Patients will receive the albumin-bound formulation of docetaxel

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤75 years, no gender limitation；
2. Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors, for which standard therapy either does not exist or has proven to be ineffective, intolerable or unacceptable for the patient；
3. At least one measurable lesion as per RECIST version 1.1；
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1；
5. Life expectancy ≥3 months；
6. Adequate bone marrow, cardiac, liver and renal function；

Exclusion Criteria:

1. Chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor treatment within 4 weeks of the first dose of the study drug, 6 weeks for mitomycin C or nitrosoureas, 2 weeks (or 5 half-lives whichever is longer) for using fluorouracil or small molecule targeted drugs, 2 weeks for using traditional Chinese medicine with anti-tumor indications；
2. Currently enrolled in any other clinical study, or administration of other investigational agents w

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced AE during cycle1. | 21 days.
  AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol specified procedure, whether or not considered related to the medicinal product/protocol specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE.
Number of participants who experienced DLT during cycle1. | 21 days.
  A DLT was graded using the National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.02 and defined as any of the following: grade 3 or 4 non-hematologic adverse events unless they were not optimally treated with supportive care; grade 3 or 4 asymptomatic laboratory abnormal values lasting >7 days; prolonged grade 2 toxicity (lasting more than 2 weeks) leading to treatment interruption and/or dose reduction; pancytopenia with a hypocellular bone marrow and no marrow blasts lasting ≥6 weeks (AL participants); grade 3 neutropenia with fever or infection (OHM participants); grade 3 thrombocytopenia with bleeding (OHM participants); or grade 4 neutropenia or thrombocytopenia, regardless of symptoms and lasting ≥3 days (OHM participants).
Classic 3+3 design to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) | Through study completion, an average of 1 year.
  The maximum tolerated dose (MTD) (if available) and recommended Phase 2 dose (RP2D) of Albumin-bound Docetaxel.

SECONDARY OUTCOMES:
Area under the concentration-time curve of Albumin-bound Docetaxel from time 0 to last (AUC 0-∞) | 21 days.
  The pharmacokinetic parameters AUC0-last of Albumin-bound Docetaxel.
Area under the concentration-time curve of Albumin-bound Docetaxel from time 0 to infinity (AUC 0-∞) | 21 days.
  The pharmacokinetic parameters AUC0-∞ of Albumin-bound Docetaxel.
Observed maximum concentration (Cmax )of Albumin-bound Docetaxel | 21 days.
  The pharmacokinetic parameters Cmax of Albumin-bound Docetaxel.
Time to maximum concentration (Tmax) of Albumin-bound Docetaxel | 21 days.
  The pharmacokinetic parameters Tmax of Albumin-bound Docetaxel.
Apparent terminal Half-Life (t1/2) of Albumin-bound Docetaxel | 21 days.
  The pharmacokinetic parameters t½ of Albumin-bound Docetaxel.
Apparent total body clearance (CL/F) of Albumin-bound Docetaxel | 21 days.
  The pharmacokinetic parameters CL/F of Albumin-bound Docetaxel.
Objective response rate (ORR) | Through study completion, an average of 1 year.
  Efficacy measures overall response rate (ORR) of Albumin-bound Docetaxel.
Progression free survival (PFS) | Through study completion, an average of 1 year.
  Efficacy measures progression-free survival (PFS) of Albumin-bound Docetaxel.
Disease control rate (DCR) | Through study completion, an average of 1 year.
  Efficacy measures disease control rate (DCR) of Albumin-bound Docetaxel.
Duration of response (DOR) | Through study completion, an average of 1 year.
  Efficacy measures duration of response (DOR) of Albumin-bound Docetaxel.

OTHER OUTCOMES:
Biomarkers of Albumin-bound Docetaxel. | 21 days.
  The correlation between the AAG level(in plasma) and albumin-bound docetaxel.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided